CLINICAL TRIAL: NCT07217886
Title: A Phase 1, Multicenter, Nonrandomized, Open-label, Parallel-group Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of S-892216-PO in Participants With Varying Degrees of Renal Impairment and Matched Control Participants With Normal Renal Function
Brief Title: A Study of S-892216-PO in Participants With Renal Impairment and Matched Controls
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2420T1614
Record Dates: First submitted 2025-10-14; First posted 2025-10-20 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Renal Impairment
Keywords: S-892216; Hemodialysis; Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A (Severe Renal Impairment) (Experimental): Participants with severe renal impairment not on HD will receive S-892216-PO.
  Interventions: Drug: S-892216-PO
- Group B (Renal Impairment) (Experimental): Participants with renal impairment requiring HD will receive S-892216-PO.
  Interventions: Drug: S-892216-PO
- Group C (Normal Renal Function) (Experimental): Participants with normal renal function will receive S-892216-PO.
  Interventions: Drug: S-892216-PO
- Group D (Moderate Renal Impairment) (Experimental): Participants with moderate impairment will receive S-892216-PO.
  Interventions: Drug: S-892216-PO
- Group D (Mild Renal Impairment) (Experimental): Participants with mild impairment will receive S-892216-PO.
  Interventions: Drug: S-892216-PO

INTERVENTIONS:
Drug: S-892216-PO — S-892216-PO tablet will be administered orally.

SUMMARY:
The purpose of this study is to measure the pharmacokinetics, safety, and tolerability of S-892216 (S-892216-PO) in participants with mild, moderate, or severe renal impairment not on dialysis, or renal impairment requiring hemodialysis (HD), and in participants with normal renal function.

ELIGIBILITY:
Key Inclusion Criteria:

* Considered to be healthy (for normal renal function participants) or medically stable (for participants with renal impairment), as determined by medical evaluation including medical history, physical examination, clinical laboratory tests, vital sign measurements, and 12-lead electrocardiogram during the screening period and on Day -1.
* Participants With Severe, Moderate, and Mild Renal Impairment not on HD (Group A, D and E): Participants that are not undergoing HD and have mild, moderate, or severe renal impairment based upon the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine formula (estimated glomerular filtration rate [eGFR]) and the participant's body surface area (BSA) calculated at the screening visit.
* Participants With Renal Impairment Requiring HD (Group B): Receiving stable HD at least 3 times a week for at least 6 months prior to screening
* Participants With Normal Renal Function: Participants with clinical laboratory tests within normal reference range for the laboratory, or abnormal but considered not clinically significant by the investigator. Renal function, calculated by the 2021 CKD-EPI creatinine formula and the participant's BSA, must be normal (that is, eGFR ≥90 milliliters/minute).

Key Exclusion Criteria:

* Participants with life expectancy less than or equal to 3 months.
* History or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, constituting a risk when taking the study intervention, or interfering with the interpretation of data based on the judgment of the investigator.
* Participants With Normal Renal Function: History or presence of renal disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, constituting a risk when taking the study intervention, or interfering with the interpretation of data.
* Participants With Any Renal Impairment (Groups A, B, D, and E): Participant with clinically significant laboratory values in the opinion of the investigator or outside protocol-specified ranges or limits during the screening period or on Day -1.
* Participants With Severe, Moderate, Mild Renal Impairment not on HD (Groups A, D, and E): Current or anticipated need for HD during the study.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of S-892216 | Day 1 (predose up to 504 hours postdose) and Day 29 (predose up to 72 hours postdose) for Group B participants only
Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration After Dosing (AUC0-last) of S-892216 | Day 1 (predose up to 504 hours postdose) and Day 29 (predose up to 72 hours postdose) for Group B participants only
Group B Only: Cumulative Amount of the Drug Recovered in Dialysate (AHD) of S-892216 | Day 1 (up to 6 hours postdose)
Group B Only: Area Under the Dialysate Concentration in the Arterial Sides of Port-time Curve During Hemodialysis (AUChd) of S-892216 | Day 1 (up to 6 hours postdose)

SECONDARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Day 1 through Day 39

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Orlando Clicinal Research Center, Orlando, Florida
  - Global Clinical Professionals (GCP) LLC, St. Petersburg, Florida
  - Genesis Clinical Research, Tampa, Florida
  - Alliance for Multispecialty Research (AMR)-Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No